CLINICAL TRIAL: NCT06922175
Title: Retrospective Evaluation of Cenobamate's Health Care Resources Utilization (HCRU) in the Management of Uncontrolled Focal Onset Seizures- A Retrospective, Chart Review Study
Brief Title: REACH: RWE Retrospective Study to Evaluate Cenobamate Impact on Health Care Resource Utilization
Status: Recruiting | Type: Observational
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: 1Med (Other)
Responsible Party: Sponsor
Other Study IDs: 169(A)AV23432
Record Dates: First submitted 2025-04-01; First posted 2025-04-10 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Epilepsy With Uncontrolled Focal-onset Seizures
Keywords: anti-seizure medications; Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adult patients affected by epilepsy with focal-onset seizures: Adult patients affected by epilepsy with focal-onset seizures not adequately controlled after 2 or more ASMs (anti-seizure medications), due to efficacy or tolerability issues, who start a treatment with cenobamate as an adjunctive therapy (according to SmPC), in real world setting, and have at least 6 months of data on treatment and HCRU (if any) prior to cenobamate starting date.

SUMMARY:
The Study is an observational, retrospective study which aim is to assess cenobamate's healthcare resources utilization (HCRU) in the management of uncontrolled focal onset seizures. The amin objective is to compare the resource utilization before and after the use of cenobamate. Data from medical charts will be used and inserted into the eCRF from which the analyses will be conducted. Data from 200 patients from 10 sites in 5 countries are included.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients of any ethnic origin ≥18 years old at index date;
2. Patients with a diagnosis of epilepsy with uncontrolled focal-onset seizures despite the previous treatment with from 2 to 5 ASMs who started treatment with cenobamate at index date;
3. Patients presenting at least 1 seizure a month in the last 6 months prior to index date;
4. Patients with at least 6 months of data coverage in the medical records prior to the index date;
5. Patients with at least 12 months of data in the medical records after index date (with a maximum interval between data of 6 months).
6. Patients who give the consent to the processing of personal data according to the General Data Protection Regulation (GDPR) and/or other applicable local regulation.

Exclusion Criteria:

1. Patients who meet any of the contraindications to the administration of adjunctive ASMs according to their approved SmPC;
2. Patients who started cenobamate within an EAP;
3. Progressive neurological disease, including degenerative CNS diseases and/or progressive brain tumors;
4. Patients with specific syndrome (e.g. LGS and Dravet);
5. Pregnancy or lactation;
6. Patients without self-judgement ability;
7. Patients with substance and alcohol abuse or dependence (except for caffeine and nicotine);
8. Patients participating in any pharmacological or nonpharmacological interventional study starting from 6 months before the index date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients affected by epilepsy with focal-onset seizures not adequately controlled after 2 or more anti-seizure medications (ASMs), due to efficacy or tolerability issues, who start a treatment with cenobamate as an adjunctive therapy (according to SmPC), in real world setting, and have at least 6 months of data on treatment and healthcare resources utilization (HCRU) (if any) prior to cenobamate starting date.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Impact of cenobamate used as adjunctive therapy on epilepsy-related healthcare resources utilization (HCRU), stratified by early and later treatment lines. | 0-12 months
  To assess the impact of cenobamate used as adjunctive therapy on epilepsy-related HCRU, will be collected the number of epilepsy/epilepsy treatment-related hospitalizations during all the observation period
Impact of cenobamate used as adjunctive therapy on epilepsy-related healthcare resources utilization (HCRU), stratified by early and later treatment lines. | 0-12 months
  To assess the impact of cenobamate used as adjunctive therapy on epilepsy-related HCRU,will be collected the length of epilepsy/epilepsy treatment-related hospitalizations during all the observation period
Impact of cenobamate used as adjunctive therapy on epilepsy-related healthcare resources utilization (HCRU), stratified by early and later treatment lines | 0-12 months
  To assess the impact of cenobamate used as adjunctive therapy on epilepsy-related HCRU will be collected the number of epilepsy/epilepsy treatment-related outpatient visits (OP) during all the observation period
Impact of cenobamate used as adjunctive therapy on epilepsy-related healthcare resources utilization (HCRU), stratified by early and later treatment lines | 0-12 months
  To assess the impact of cenobamate used as adjunctive therapy on epilepsy-related HCRU will be collected the number of epilepsy/epilepsy treatment-related emergency room (ER) visits;

SECONDARY OUTCOMES:
Impact of cenobamate used as adjunctive therapy on the use of concomitant anti-seizure medications (ASMs) | 0-12 months
  To assess the impact of cenobamate used as adjunctive therapy on the use of concomitant anti-seizure medications (ASMs), the following data will be recorded: Switch/add-on of other ASMs
Impact of cenobamate used as adjunctive therapy on the use of concomitant anti-seizure medications (ASMs) | 0-12 months
  To assess the impact of cenobamate used as adjunctive therapy on the use of concomitant anti-seizure medications (ASMs), the following data will be recorded: Changes in the dose of co-ASMs
Impact of cenobamate used as adjunctive therapy on the use of concomitant anti-seizure medications (ASMs) | 0-12 months
  To assess the impact of cenobamate used as adjunctive therapy on the use of concomitant anti-seizure medications (ASMs), the following data will be recorded: Changes in the number of co-ASMs
Impact of cenobamate used as adjunctive therapy on the use of concomitant anti-seizure medications (ASMs) | 0-12 months
  To assess the impact of cenobamate used as adjunctive therapy on the use of concomitant anti-seizure medications (ASMs), the following data will be recorded: Time to discontinuation of ASMs
Impact of cenobamate used as adjunctive therapy on epilepsy-related emergency and medical care | 0-12 months
  To evaluate the impact of cenobamate used as adjunctive therapy on epilepsy-related emergency and medical care, the number of epilepsy/epilepsy treatment related emergency care, ambulance use, the number of outpatient visits with neurologists, and the number of epilepsy specialist nurses' intervention will be collected;
Effectiveness of cenobamate used as adjunctive therapy | 0-12 months
  To evaluate the effectiveness of cenobamate used as adjunctive therapy, seizure frequency at baseline and at routinely scheduled follow-up visits, till the end of observation will be collected. For comparability, seizure frequency will be extrapolated per month (28 days);
Impact of cenobamate used as adjunctive therapy on epilepsy-related surgery | 0-12 months
  To assess the impact of cenobamate used as adjunctive therapy on epilepsy-related surgery the following data will be collected:
  * the number of epilepsy-related surgery (how many patients initiated cenobamate while they were in waiting list or post-surgical intervention, i.e. surgical failure);
  * the number of hospitalizations due to surgery related to epilepsy (e.g. fractures due to falls);
  * the number of Intensive Care Unit (ICU) visits;
Impact of cenobamate used as adjunctive therapy on comorbidity-related healthcare resources utilization (HCRU) | 0-12 months
  To evaluate the impact of cenobamate used as adjunctive therapy on comorbidity-related HCRU, the following data will be collected:
  * Number and length of hospitalizations of all-cause inpatient visits,
  * Number of ER visits,
  * Number of outpatient visits. All-cause HCRU will be defined as HCRU due to any cause;
Impact of cenobamate used as adjunctive therapy on phone calls/virtual interventions | 0-12 months
  To evaluate the impact of cenobamate used as adjunctive therapy on phone calls/virtual interventions, the number of phone calls/virtual interventions will be collected.
Safety of cenobamate used as adjunctive therapy | 0-12 months
  To evaluate safety of cenobamate used as adjunctive therapy, the number, type and severity of, adverse events, adverse drug reactions will be collected. Moreover, changes in the number, type, dose of concomitant medications other than anti-seizure medications will be collected over the duration of the study.

CONTACTS AND LOCATIONS:
Locations (10):
- Germany (3):
  - Epilepsiezentrums am Neurozentrum des Universitätsklinikum Freiburg, Freiburg im Breisgau, Germany
  - Epileptologicum, Hamburg, Germany
  - Diakonie Kork, Epilepsiezentrum, Kork, Germany
- Kempenhaeghe - Academisch Centrum voor Epilepsie, Heeze, Netherlands, Netherlands
- Spain (3):
  - Epilepsy Unit - Neurology Department Valle de Hebron Hospital, Barcelona, Spain
  - Epilepsy Unit of the Neurology Department of the Hospital Clínico San Carlos, Madrid, Spain
  - Consorcio Hosp. General Universitario Valencia, Valencia, Spain
- Department of Neurology, University Hospital Zurich, Zurich, Switzerland, Switzerland
- United Kingdom (2):
  - Institute of Neurosciences NHS Greater Glasgow and Clyde, Glasgow, UK
  - Epilepsies - The Royal Wolverhampton NHS Trust, Wolverhampton, UK